CLINICAL TRIAL: NCT01167530
Title: Study to Evaluate RAD001 in Combination With Radiotherapy in Non-small Cell Lung Cancer
Acronym: RAD001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGR 1269
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2010-07

CONDITIONS: Non-small Cell Lung Cancer; Locally Advanced Disease
Keywords: Everolimus; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Everolimus — First phase of the study:RAD001 (everolimus) will be administered per os every Monday, one week before then during the radiotherapy and will be continued for 3.5 weeks after the end of the radiotherapy. Chemotherapy is given 4.5 weeks after the end of radiotherapy. Three patient cohorts are planned, receiving 10, 20 and 50 mg of RAD001 per week.Second phase of the study:RAD001 (everolimus) will be administered per os every day one week before then during the radiotherapy and will be continued for 3.5 weeks after the end of radiotherapy. Chemotherapy is given 4.5 weeks after the end of radiotherapy. Three patient cohorts are planned, receiving 2.5, 5 and 10 mg of RAD001 per day.The two phases of the study may be conducted independently and in parallel.

SUMMARY:
The phase 1 study evaluats RAD001 in combination with radiotherapy in non-small cell lung cancer.

First phase of the study:RAD001 (everolimus) will be administered per os every Monday, one week before then during the radiotherapy and will be continued for 3.5 weeks after the end of the radiotherapy. Chemotherapy is given 4.5 weeks after the end of radiotherapy. Three patient cohorts are planned, receiving 10, 20 and 50 mg of RAD001 per week.Second phase of the study:RAD001 (everolimus) will be administered per os every day one week before then during the radiotherapy and will be continued for 3.5 weeks after the end of radiotherapy. Chemotherapy is given 4.5 weeks after the end of radiotherapy. Three patient cohorts are planned, receiving 2.5, 5 and 10 mg of RAD001 per day.The two phases of the study may be conducted independently and in parallel.Radiotherapy: 66 Grays over 6.5 weeks. (5 weekly fractions of 2 Grays)Chemotherapy: 2 cycles: Cisplatin 100 mg/m2 D1, Navelbine 25 mg/m2 D1, D8, every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable non-small cell lung cancer, stage IIIA/B, or stage IV for which the primary tumor is symptomatic (cough, dyspnea, pain) without extra-thoracic lesions rapidly evolving for which patients should receive radiotherapy at curative dose
2. Measurable lesion, documented histologically, potentially accessible during fiberoptic bronchoscopy.
3. Age > 18 years, WHO 0-1,
4. Neutrophil count > 1500 /mm3, Hemoglobin > 9 g/dL, Platelet count > 100,000/mm3
5. Bilirubin < 1.5 mg/dL, Transaminases < 3 N, albumin >30 g / L, PT > 70%
6. Creatinine < 120 μM/L
7. Patient information and informed consent form signed.
8. No previous treatment for lung cancer (surgery, radiotherapy, chemotherapy).

Exclusion Criteria:

1. Patients previously treated with RAD001 (everolimus) or any other mTOR inhibitor
2. Stage IV for which the primary tumor is not symptomatic with extra-thoracic lesions rapidly evolving requiring systemic treatment
3. Previous radiotherapy,
4. Venous or arterial thrombosis, pulmonary embolism during the previous six months
5. Concomitant treatment with phenytoin, phenobarbital or any other antiepileptic agent, history of epilepsy
6. Concomitant treatment with medicinal products that inhibit, induce or are substrates for CYP3A4(inhibitors: atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, amprenavir, aprepitant, diltiazem, erythromycin, fluconazole, fosamprenavir, verapamil, ciclosporin, voriconazoleinducers: rifampicin, carbamazepine, rifabutinsubstrates: midazolam, buspirone, felodipine)
7. Concomitant therapy with agents otherwise used in the treatment of cancer (for example methotrexate for rheumatoid arthritis).
8. Chronic treatment with corticosteroids or another immunosuppressant
9. Patients with an active bleeding diathesis or taking an oral vitamin K antagonist (except low-dose Coumadin (warfarin sodium))
10. Other concurrent severe and/or uncontrolled disease which could compromise participation in the study (i.e. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, unstable angina, or congestive heart failure - New York Heart Association Class III or IV, ventricular arrhythmia, active ischemic heart disease, myocardial infarction during the previous six months, chronic liver or renal disease, active upper GI tract ulceration)
11. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (EVEROLIMUS) (i.e. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
12. HIV seropositivity
13. Patient with a virological test positive to hepatitis B (HBs positive)
14. Patients with active cutaneous, mucosal, ocular or gastrointestinal disorders of grade > 1
15. Previous cancer (except basal cell skin cancer or cervical carcinoma in situ) during the 3 years prior to entering the trial.
16. important pulmonary fibrosis on X-ray
17. Women who are or could become pregnant or who are currently breastfeeding,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-03; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Toxicity | Eleven week
  Dose limiting toxicity

SECONDARY OUTCOMES:
Progression-free and overall survival. | Three years
Response rate | Four months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- See also: Related Info — http://www.igr.fr/